CLINICAL TRIAL: NCT06176976
Title: Preoperative Administration of Lugols Solution in Toxic Thyroid Diseases (TD): A Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Styliani Konstantinos Laskou, Principal Investigator, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LS trial
Record Dates: First submitted 2023-11-29; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Toxic; Thyroid
MeSH Terms: conditions — Thyrotoxicosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thyroidectomy without lugols solution preparation (No Intervention): euthyroid patients undergoing total thyroidectomy for toxic thyroid disease, no preoperative preparation with 5% lugols solution
- Thyroidectomy with lugols solution preparation (Experimental): euthyroid patients undergoing total thyroidectomy for toxic thyroid disease, preoperative preparation with 5% lugols solution for 10 days
  Interventions: Dietary Supplement: Lugol's iodine solution 5%

INTERVENTIONS:
Dietary Supplement: Lugol's iodine solution 5% — 4 drops of LS every 8 hours for 10 days preoperatively will be given
  Arms: Thyroidectomy with lugols solution preparation

SUMMARY:
Lugol's solution and other preparations containing iodide have been used as an adjuvant treatment in patients with toxic disease planned for thyroidectomy. However, no conclusive evidence supporting the benefits of preoperative treatment with LS for patients with toxic goiters. This trial aims to provide new insights into future recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age
* Toxic thyroid disease, treated with antithyroid drugs, euthyroid and proposed for total thyroidectomy
* Written informed consent

Exclusion Criteria:

* prior thyroid or parathyroid surgery,
* hyperparathyroidism that requires associated parathyroidectomy,
* thyroid cancer that requires adding a lymph node dissection,
* iodine allergy,
* consumption of lithium or amiodarone,
* medically unfit patients (ASA-IV),
* breastfeeding women,
* preoperative vocal cord palsy and
* planned endoscopic, video-assisted or remote access surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Thyroidectomy complications rate | 24 hours postoperatively
  postoperative bleeding, hypoparathyroidism and recurrent laryngeal nerve palsy will be recorded

SECONDARY OUTCOMES:
Thyroid volume | Pre-intervention and immediately after the intervention for the lugols solution group. Only preoperative measurement for the non lugols solutiongroup.
  via ultrasound
Superior thyroid artery blood flow | Pre-intervention and immediately after the intervention for the lugols solution group. Only preoperative measurement for the non lugols solutiongroup.
  via ultrasound
Fibrinogen | Pre-intervention and immediately after the intervention for the lugols solution group. Only preoperative measurement for the non lugols solutiongroup.
  Sera, stored at -80 C until they were used
Vascular endothelial growth factor | Pre-intervention and immediately after the intervention for the lugols solution group. Only preoperative measurement for the non lugols solutiongroup.
  Sera, stored at -80 C until they were used
Interleukin-16 serum levels | Pre-intervention and immediately after the intervention for the lugols solution group. Only preoperative measurement for the non lugols solutiongroup.
  Sera, stored at -80 C until they were used
Thromboelastography | Pre-intervention and immediately after the intervention for the lugols solution group. Only preoperative measurement for the non lugols solutiongroup.
  Thromboelastography assay

CONTACTS AND LOCATIONS:
Overall Officials: Styliani Laskou, Principal Investigator — 3rd Surgical Department of Aristotle University, AHEPA University Hospital, Thessaloniki
Locations (1):
- 3rd Surgical Department of Aristotle University, AHEPA University Hospital, Thessaloniki, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No